CLINICAL TRIAL: NCT04658693
Title: Functional and Neuroprotective Effects of Restoring Lower Limb Sensation After Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: A3566-R; 1583890 (Other: IRBnet); RX003566-01A1 (Other Grant/Funding Number: VA Rehabilitation R&D)
Record Dates: First submitted 2020-11-20; First posted 2020-12-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lower Extremity Amputee; Diabetic Peripheral Neuropathy
Keywords: Sensory Feedback; Limb Loss; Prosthesis User

STUDY DESIGN:
Intervention Model Description: The project will take the form of a series of controlled single-subject feasibility and proof-of-concept studies with repeated measures. Subjects will act as their own concurrent controls with and without sensory stimulation, as well as their own longitudinal (historical) controls pre- and post-implementation of the Sensory Neuroprosthesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Multi contact electrode implant and implanted electromyography recording electrodes (Experimental): Fifteen subjects with lower limb amputation will receive implanted multicontact stimulating nerve cuff electrodes connected to temporary percutaneous leads.
  During experimental testing, a small amount of stimulation will be applied to the nerves through the contacts of the multichannel cuff electrode.
  Interventions: Device: Implanted Multi contact stimulating electrode and intramuscular electromyography recording electrode

INTERVENTIONS:
Device: Implanted Multi contact stimulating electrode and intramuscular electromyography recording electrode — See arm description
  Other Names: Sensory Neuroprosthesis

SUMMARY:
The purpose of this study is to evaluate the effectiveness of providing sensation of the missing limb to individuals with above and below the knee limb loss. The investigators will implanted stimulating electrodes to send small electrical currents to the remaining nerves. These small electrical currents cause the nerves to generate signals that are then transferred to your brain similar to how the information about your foot and lower limb used to be transferred to the brain prior to your limb loss. Additionally, there is the option to have muscle recording electrodes implanted within the muscles of the lower limb with the goal to develop a motor controller that would allow the user to have intuitive control of a robotic prosthetic leg.

DETAILED DESCRIPTION:
Electrodes are surgically implanted on one to four nerves of the residual limb. Intramuscular recording electrodes can be implanted in the lower limbs and hip muscles in order to obtain electromyography (EMG) signals. The EMG recordings will be used to develop an algorithm which can operate an advanced robotic prosthesis in which the prosthesis joint(s) movements could be controlled. An external wearable stimulation device controls the delivery of electrical pulses to the implanted system. An instrumented prosthesis will be developed such that perceived sensations would correspond to prosthesis interactions with the floor. The instrumented prosthesis will be worn while the participant is engaging in various functional tasks, such as standing, walking or climbing stairs or with visual or mental distractions.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, medically stable lower limb amputation due to diabetes or insensate foot due to Diabetic peripheral neuropathy
* Being ambulatory and ability to stand or walk with prosthesis or orthosis
* Viable target nerves in the lower extremity as determined by standard-of-care clinical tests of nerve conduction, response to stimulation, sensory evoked potentials (SEP) and the like
* Good skin integrity and personal hygiene
* Absence of autoimmune deficiencies, seizure disorders or cardiac abnormalities contraindicating stimulation
* Sufficient social support and personal ability to tolerate study procedures and comply with follow-up schedule

Exclusion Criteria:

* Active pressure ulcers or chronic skin ulcerations
* Uncontrolled diabetes with HbA1c greater than or equal to 69 mmol/mol (8.5%)
* Significant vascular disease
* Significant history of poor wound healing
* Significant history of uncontrolled infections
* Active infection
* Significant pain in the foot, residual or phantom limb
* Pregnancy
* Inability to speak English: The study design requires the subject to communicate and describe the elicited sensations in their lower limb
* History of vestibular or movement disorders that would compromise balance or walking
* Class II or III obesity (Body Mass Index > 35)
* Uncontrolled depression, psychoses or cognitive impairments. Subjects with unstable mental illness or severe cognitive impairments may be unable to comply with a long term study schedule
* Expectation that MRI will be required at any point for the duration of study or while percutaneous leads are in place. At this time MRI is contraindicated, subjects who require regular MRI should not enroll
* Arthritis in the area of implant- Inflammation or stiffness in the area of implant could limit placement of the electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2027-09-02 (Estimated); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
Stimulation thresholds | 9 months post implant
  Quantify the minimum stimulation required to evoke electrically induced sensations on the phantom limb.
Functional Gait Assessment (FGA) | 6 months post implant
  The Functional Gait Assessment is a 10 task test that measures postural stability. Each task is scored from 0 -3 with 0 indicating severe impairment in the task and 3 indicating normal ambulation. The scores are combined to give a total score. The maximum score is 30. A higher score indicates a better outcome.

SECONDARY OUTCOMES:
Neuropathic Pain Syndrome Inventory (NPSI) | 4 years post implant
  The NPSI is comprised of five subscales, each representing different dimensions of neuropathic pain: burning spontaneous pain (burning), pressing spontaneous pain (pressing), paroxysmal pain (paroxysmal), evoked pain (evoked), and paresthesia/dysesthesia Each area subscale is scored between 0-10. The scores are not combined, but are able to report on different aspects of neuropathic pain. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Triolo, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be provided upon request.

REFERENCES:
- See also: VA Center of Excellence website listing this and other ongoing studies. — https://www.aptcenter.research.va.gov/